CLINICAL TRIAL: NCT01895946
Title: A Phase I, Open-Label, Multicentre Study to Compare Two Dosage Formulations of AZD5363 and to Establish the Effect of Food on the Pharmacokinetic Exposure, Safety and Tolerability of AZD5363 in Patients With Advanced Solid Malignancies
Brief Title: Comparison of Two Formulations of AZD5363 and the Effect of Food on Pharmacokinetic Exposure, Safety and Tolerability
Acronym: OAK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3610C00007
Record Dates: First submitted 2013-06-21; First posted 2013-07-11 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Advanced Solid Malignancy,; Safety and Tolerability,; Pharmacokinetics, Pharmacodynamics,; Tumour Response,
Keywords: Advanced solid malignancy, AZD5363,; food effect,; formulation comparison
MeSH Terms: interventions — capivasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A: Formulation Switch (Experimental): AZD5363 tablet twice daily followed by AZD5363 capsule twice daily on an intermittent regimen (4 days on, 3 days off).
  Interventions: Drug: AZD5363
- Part B: Food effect (Experimental): AZD5363 tablet twice daily on an intermittent regimen (4 days on, 3 days off) with/without food on one occasion
  Interventions: Drug: AZD5363

INTERVENTIONS:
Drug: AZD5363 — Oral AZD5363 twice daily, 4 days on 3 days off: tablet formulation for one week, followed by two weeks with capsule formulation.
  Arms: Part A: Formulation Switch
Drug: AZD5363 — Oral AZD5363 twice daily, 4 days on 3 days off, tablet formulation. On day 4 AZD5363 tablet without food. On day 11 AZD5363 tablet with food.
  Arms: Part B: Food effect

SUMMARY:
Comparison of Two Formulations of AZD5363 and the Effect of Food on Pharmacokinetic Exposure, Safety and Tolerability

DETAILED DESCRIPTION:
This study is designed to investigate the safety, tolerability and pharmacokinetics of a new drug, AZD5363, in patients with advanced cancer . This study will investigate how the body handles AZD5363 (ie, how quickly the body absorbs and removes the drug), the comparison of a capsule and a tablet formulation and the effect of food on AZD5363 tablet formulation.

ELIGIBILITY:
Inclusion Criteria: -

* Aged at least 18 years
* The presence of a solid, malignant tumour, excluding lymphoma, that is resistance to standard therapies or for which no standard therapies exist
* The presence of at least one lesion that can be accurately assessed at baseline by Computerised Tomography (CT), Magnetic Resonance Imaging (MRI) or plain X-ray and is suitable for repeated assessment
* Estimated life expectancy of more than 12 weeks

Exclusion Criteria: -

* Clinically significant abnormalities of glucose metabolism
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable (not requiring steroids)
* Evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses or active infections including hepatitis B, C and Human Immunodeficiency Virus (HIV)
* Evidence of clinically significant cardiac abnormalities, uncontrolled hypotension, left ventricular ejection fraction below the lower limit of normal for the site or experience of significant cardiac interventional procedures
* A bad reaction to AZD5363 or any drugs similar to it in structure or class

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Lindemann, MSD, Study Director — AstraZeneca; Udai Banerji, MD, PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (3):
- Research Site, Amsterdam, Netherlands
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Surrey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 parts to this study: Part A (tablet formulation assessment) followed by Part B (food effect assessment). Part A: first patient enrolled on 18/12/2013 and last patient completed on 16/12/2014. Part B: first patient enrolled on 10/09/2014 and last patient completed on 22/07/2015. Part A was conducted at 3 sites and Part B at 2 sites.
Pre-assignment Details: Note, Part A involved a cross over between tablet and capsule formulations A total of 33 patients were enrolled. 30 of these patients passed screening assessments and were dosed
Groups:
- Part A: Part A of the study
- Part B: Part B of the study
Period: Overall Study
Arm/Group | Part A | Part B
Started | 18 | 12
Completed | 18 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 18 | 12 | 30
Age, Customized [Number; unit: Participants] — Age group, customized
  Participants
    <50 years | 4 | 1 | 5
    Between 50 and 65 years | 9 | 6 | 15
    >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Gender, Male/Femelle
  Participants
    Female | 8 | 7 | 15
    Male | 10 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Ratio of Css,Max for Day 4 to Day 11
Description: The actual sampling times were used in the pharmacokinetics (PK) parameter calculations and PK parameters were derived using standard non-compartmental methods.
  Following the twice daily dosing in Cycle 1 at Day 4 and 11 for both the formulation switch and food effect investigations, the following PK parameters have been determined:
  Maximum plasma concentration at steady state (Css max), time to Css,max (tss max), minimum plasma concentration at steady state (Css min), area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCss) and apparent clearance (CLss/F).
  Css max, tss max were determined by inspection of the concentration-time profiles. AUCss was calculated using the linear up / log down trapezoidal rule. CLss/F was determined from the ratio of dose/AUCss.
  Ratio of Css,max for Day 4 to Day 11 have been derived.
Time Frame: Day 4 and Day 11
Population: All patients who provided concentration-time data for AZD5363 for both capsule and tablet administration (Part A) or for both fed and fasted treatments and who were compliant with the standard dietary and evaluability requirements (Part B) were included in PK analysis set.
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Part A | Part B
Number analyzed (Participants) | 11 | 9
Ratio | 1.02 [0.86 to 1.20] | 0.67 [0.55 to 0.82]
Statistical Analysis 1: Comparison: Part A; Test type: Superiority or Other; Mixed Models Analysis; Least square mean difference (LSM) = 1.02, 90% CI 2-sided [0.86 to 1.20]
Statistical Analysis 2: Comparison: Part B; Test type: Superiority or Other; Mixed Models Analysis; Least square means difference (LSM) = 0.67, 90% CI 2-sided [0.55 to 0.82]

2. Primary Outcome: Ratio of AUCss for Day 4 to Day 11
Description: The actual sampling times were used in the parameter calculations and PK parameters were derived using standard non-compartmental methods.
  Following the twice daily dosing in Cycle 1 at Day 4 and 11 for both the formulation switch and food effect investigations, the following PK parameters have been determined:
  Css max, tss max, Css min, area under the plasma concentration-time curve from zero to the end of the dosing interval (AUCss) and CLss/F.
  Css max, tss max were determined by inspection of the concentration-time profiles. AUCss was calculated using the linear up / log down trapezoidal rule. CLss/F was determined from the ratio of dose/AUCss.
  Ratio of AUCss for Day 4 to Day 11 have been derived.
Time Frame: Day 4 and Day 11
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Part A | Part B
Number analyzed (Participants) | 11 | 9
Ratio | 0.90 [0.77 to 1.06] | 0.89 [0.76 to 1.05]
Statistical Analysis 1: Comparison: Part A; Test type: Superiority or Other; Mixed Models Analysis; Least square means difference (LSM) = 0.90, 90% CI 2-sided [0.77 to 1.06]
Statistical Analysis 2: Comparison: Part B; Test type: Superiority or Other; Mixed Models Analysis; Least square means difference (LSM) = 0.89, 90% CI 2-sided [0.76 to 1.05]

3. Secondary Outcome: Efficacy: Best Objective Response (BOR)
Description: Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 guidelines for measurable, non-measurable, target lesions (TLs) and non-target lesions (NTLs) and the objective tumour response criteria was used.
  Categorisation of objective tumour response assessment was based on the RECIST 1.1 guidelines for response: CR (complete response, efined as disappearance of all target lesions), PR (partial response, defined as >=30% decrease in the sum of the longest diameter of target lesions), SD (stable disease, defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression) and PD (progression of disease, defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion). BOR was the best overall response observed across the study and up to 36 weeks. Number of subjects with response (CR or PR) is described.
Time Frame: Assessed every 6 weeks, up to 36 weeks
Population: Modified intent-to-treat analysis set: all patients who received at least one dose of study treatment with a baseline tumour assessment.
Measure: Number; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 18 | 12
Participants | 0 | 0

4. Secondary Outcome: Efficacy: Disease Control at Week 12
Description: Disease control = confirmed complete response + confirmed partial response + stable disease at 12 weeks
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Part A | Part B
Number analyzed (Participants) | 18 | 12
Participants | 1 | 3

5. Secondary Outcome: Efficacy: Target Lesion Size, Percentage Change From Baseline at Week 12
Description: Tumour size is the sum of the longest diameters of the target lesions. Target lesions are measurable tumour lesions.
  The percentage change in target lesion tumour size at each week 12 for which data are available was obtained for each subject taking the difference between the sum of the target lesion at each week 12 and the sum of the target lesions at baseline divided by the sum of the target lesions at baseline multiplied by 100 (i.e. (week 12) - baseline)/baseline * 100).
Time Frame: Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Part A | Part B
Number analyzed (Participants) | 6 | 7
Percentage change from baseline | 8.1 (14.72) | -1.5 (6.49)

6. Secondary Outcome: Efficacy: Target Lesion Size, Best Percentage Change From Baseline
Description: Tumour size is the sum of the longest diameters of the target lesions. Target lesions are measurable tumour lesions.
  best percentage change in tumour size from baseline is the maximum reduction from baseline or the minimum increase from baseline in the absence of a reduction from baseline based on all post baseline assessments.
Time Frame: Assessed every 6 weeks up to 36 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage change from baseline
Arm/Group | Part A | Part B
Number analyzed (Participants) | 14 | 11
Percentage change from baseline | 10.5 (13.62) | 0.2 (9.92)

7. Secondary Outcome: Efficacy: Progression-free Survival (PFS)
Description: PFS is defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the subject withdraws from randomised therapy or receives another anti-cancer therapy prior to progression. Subjects who have not progressed or died at the time of analysis were censored at the time of the latest date of assessment from their last evaluable RECIST assessment. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a nontarget lesion, or the appearance of new lesions.
Time Frame: Assessed every 6 weeks up to 36 weeks
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Part A | Part B
Number analyzed (Participants) | 18 | 12
weeks | 6.1 (13.62) [5.0 to 16.7] | 13.7 (9.92) [11.1 to 35.4]

ADVERSE EVENTS:
Time Frame: Adverse events with an onset date on or after the date of first dose and up to and including 28 days following the date of last dose of study medication were collected.
Arm/Group | Part A | Part B
Serious Adverse Events (participants affected / at risk) | 5/18 | 6/12
Other Adverse Events (participants affected / at risk) | 18/18 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=18) | Part B (N=12)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pneumonia mycoplasmal (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=18) | Part B (N=12)
Diarrhoea (Gastrointestinal disorders) | 14 (36) | 9 (14)
Fatigue (General disorders) | 7 (9) | 8 (9)
Nausea (Gastrointestinal disorders) | 8 (9) | 8 (11)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (16) | 6 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (6)
Vomiting (Gastrointestinal disorders) | 5 (9) | 5 (7)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (4)
Pyrexia (General disorders) | 2 (3) | 3 (3)
Respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (2)
Electrocardiogram QT prolonged (Investigations) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (3) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Supropubic pain (General disorders) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine decreased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Small numbers of patients in the first (fasted) and second (fed) treatment periods overall make interpretation difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No